CLINICAL TRIAL: NCT05410808
Title: Levels of Anxiety, Depression, and Quality of Life in Patients With Fibromyalgia During the COVID-19 Pandemic: A Cross-sectional Study
Brief Title: Anxiety, Depression, and Quality of Life in Patients With Fibromyalgia During the Coronavirus Disease 2019 Pandemic
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ece Cinar, Principal investigator, Ege University
Other Study IDs: 21-1T/52
Record Dates: First submitted 2022-06-05; First posted 2022-06-08 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Fibromyalgia; Coronavirus Disease 2019 Pandemic
Keywords: fibromyalgia; coronavirus disease 2019; pain; anxiety; quality of life
MeSH Terms: conditions — Fibromyalgia; COVID-19; Pain; Anxiety Disorders | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia patients: Patients diagnosed as having fibromyalgia according to the American College of Rheumatology 2016 classification criteria
  Interventions: Other: Questionnaires and physical examination
- Healthy controls: Subjects not having fibromyalgia and who live in the same household as the fibromyalgia patients
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaires and physical examination — Patients will be examined and demographic data, disease characteristics will be recorded. Health Survey Questionnaire Short Form 36 , coronavirus disease 2019 anxiety scale ,Obsession with coronavirus disease 2019 scale, and Resilience scale for adults will be answered
  Groups: Fibromyalgia patients
Other: Questionnaire — Demographic data will be recorded. Health Survey Questionnaire Short Form 36 , coronavirus disease 2019 anxiety scale ,Obsession with coronavirus disease 2019 scale, and Resilience scale for adults will be answered
  Groups: Healthy controls

SUMMARY:
Fibromyalgia patients and controls living in the same household will be evaluated for levels of resilience, covid-19 related anxiety, coronavirus disease 2019 related obsession, quality of life and pain and comparisons and correlation analyses will be carried out.

DETAILED DESCRIPTION:
Fibromyalgia is a generalized pain condition that is accompanied by sleep disturbances, anxiety, depression and somatic symptoms. During Coronavirus disease 2019 pandemic, fibromyalgia patients as well as the general population have increased anxiety levels. This study was planned to evaluate fibromyalgia patients' levels of coronavirus disease 2019 related resilience, anxiety, obsession levels about coronavirus disease 2019, quality of life and pain levels and compare them with healthy controls living in the same household.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of fibromyalgia according to the American college of rheumatology 2016 classification criteria
* Older than 18 years of age

Exclusion Criteria:

* Illiteracy
* A history of coronavirus disease 2019 infection in the last month
* Change in medication to treat fibromyalgia in the last 3 months
* Living alone (lack of a control subject)
* Severe neurological or psychiatric disorder that might hinder subjects' ability to answer the study questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with fibromyalgia and who are older than 18 years of age and controls that live in the same household as the fibromyalgia patients
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Resilience | Day 1
  Immunity against traumatic life events, measured by resilience scale for adults
Covid anxiety | Day 1
  Covid related anxiety levels, measured by covid-19 anxiety scale
Obsession with covid-19 | Day 1
  Obsession with covid-19, measured by obsession with covid scale
Quality of life assessment | Day 1
  Measured by Health Survey Questionnaire Short Form 36

CONTACTS AND LOCATIONS:
Overall Officials: Ece Cinar, MD, Principal Investigator — Principal Investigator
Locations (1):
- Ege University School of Medicine, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazza MG, De Lorenzo R, Conte C, Poletti S, Vai B, Bollettini I, Melloni EMT, Furlan R, Ciceri F, Rovere-Querini P; COVID-19 BioB Outpatient Clinic Study group; Benedetti F. Anxiety and depression in COVID-19 survivors: Role of inflammatory and clinical predictors. Brain Behav Immun. 2020 Oct;89:594-600. doi: 10.1016/j.bbi.2020.07.037. Epub 2020 Jul 30. PMID 32738287
- [Background] Qiu J, Shen B, Zhao M, Wang Z, Xie B, Xu Y. A nationwide survey of psychological distress among Chinese people in the COVID-19 epidemic: implications and policy recommendations. Gen Psychiatr. 2020 Mar 6;33(2):e100213. doi: 10.1136/gpsych-2020-100213. eCollection 2020. PMID 32215365
- [Background] Cankurtaran D, Tezel N, Ercan B, Yildiz SY, Akyuz EU. The effects of COVID-19 fear and anxiety on symptom severity, sleep quality, and mood in patients with fibromyalgia: a pilot study. Adv Rheumatol. 2021 Jun 30;61(1):41. doi: 10.1186/s42358-021-00200-9. PMID 34193303